CLINICAL TRIAL: NCT04399668
Title: Comparison of a Preoperative Ultrasound-determined and the Intraoperative #Enzian-classification in Patients With Deep Endometriosis (DE)
Brief Title: Comparison of Ultrasound-determined and Intraoperative #Enzian-classification in Patients With Deep Endometriosis
Status: Completed | Type: Observational
Sponsor: Univ.-Doz. Dr.med.univ. Gernot Hudelist, MSc. (Other)
Responsible Party: Sponsor-Investigator, Univ.-Doz. Dr.med.univ. Gernot Hudelist, MSc., MD, MSc Clinical Lecturer, Woman and Health Private Clinic Vienna
Organization: Woman and Health Private Clinic Vienna (Other)
Other Study IDs: 1
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; Deep endometriosis (DE); Transvaginal sonography (TVS); Enzian classification; #Enzian classification
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Enzian classification, which was developed in order to describe deep endometriotic (DE) lesions, is determined intraoperatively by the surgeon. Transvaginal ultrasound (TVS) examination is considered as the first-line imaging technique for endometriosis. The aim of this study is to compare the assessment of presence and severity grade of endometriotic lesions in different #Enzian compartments by a preoperative ultrasound examination to the definitive intraoperative Enzian classification using the latest revision of the Enzian classification (#Enzian).

DETAILED DESCRIPTION:
Endometriosis is a common disease with endometriotic lesions being found in the ovaries, peritoneum, or as deep endometriosis (DE) involving different pelvic organs and structures. In order to describe DE lesions, the Enzian classification was developed. In the last revision of this Enzian classification, the so-called #Enzian, presence and severity grades of ovarian and peritoneal endometriosis as well as adhesions involving tubes and ovaries are also described in addition to DE lesions.

The Enzian classification is determined intraoperatively by the surgeon. Transvaginal ultrasound (TVS) examination is considered to be the first-line imaging technique for this disease. Therefore, the aim of this study is to compare the assessment of presence and severity grade of endometriotic lesions in different #Enzian compartments by a preoperative ultrasound examination (in the form of an US-#Enzian classification) to the definitive intraoperative Enzian classification (OP-#Enzian) using the latest revision of the Enzian classification (#Enzian).

ELIGIBILITY:
Inclusion Criteria:

* All women who are scheduled for a radical surgical treatment of deep endometriosis (DE) and who undergo preoperative evaluation by transvaginal sonography (TVS)

Exclusion Criteria:

* Diagnosed or suspected malignancy
* Previous colorectal surgery or previous surgery for DE including full thickness bowel resection, vaginal resection or excision of a DE lesion involving the urinary bladder
* Virgo intacta women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who are scheduled for a radical surgical treatment of deep endometriosis (DE), undergo preoperative evaluation by transvaginal sonography (TVS) and don't fall under the exclusion criteria will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 745 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Percentages of concordances between preoperative TVS defined #Enzian with the intraoperatively determined #Enzian classification in each #Enzian compartment | 1 to 7 days
  The percentages of concordantly described endometriotic lesions including the respective lesion sizes by the preoperative TVS defined #Enzian in each #Enzian compartment will be assessed, with the intraoperatively determined #Enzian classification taken as the reference, i.e. gold standard.

SECONDARY OUTCOMES:
Sensitivity and specificity for the detection of endometriotic lesions by preoperative TVS examination using #Enzian | 1 to 7 days
  Sensitivity and specificity for the detection of endometriotic lesions in different #Enzian compartments by the preoperative TVS examination (#Enzian) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Hudelist, MD, MSc, Principal Investigator — Woman & Health Private Clinic Vienna
Locations (1):
- St. John of God Hospital Vienna, Vienna, Austria